CLINICAL TRIAL: NCT06812169
Title: The Effectiveness of USG-guided Tap Block in Postoperative Pain Relief in Pediatric Patients Who Underwent Open Appendectomy with Mc-Burney Incision
Brief Title: The Effect of Tap Block in Pain Relief in Pediatric Patients
Status: Completed | Type: Observational
Sponsor: Arnavutkoy State Hospital (Other)
Responsible Party: Principal Investigator, GOKHAN ASLAN, Specialist Anesthesiology, Arnavutkoy State Hospital
Other Study IDs: GK-TAP-GAZ
Record Dates: First submitted 2025-02-01; First posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-01

CONDITIONS: Opioid Analgesia; Pain, Postoperative; Pain Score Reduction
Keywords: TAP Block
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group S: TAP block was applied to this group of open appendectomy patients.
- Group C: TAP block was not applied to this group of open appendectomy patients.

SUMMARY:
TAP block applied for analgesic purposes in pediatric patients undergoing appendectomy surgery provides superior analgesia in analgesic relief in the first 24 hours postoperatively compared to the placebo-control group without any block. The objective of this study was to investigate the postoperative analgesic effectiveness of TAP block based on postoperative pain scores in pediatric patients undergoing appendectomy surgery. This study is valuable because of there are a limited number of studies in this field in pediatric patients in the literature.

DETAILED DESCRIPTION:
This study was designed as prospectif, randomized, placebo-controlled, double-blind. A total of 60 pediatric patients, who were planned to undergo elective open appendectomy surgery under general anesthesia, were included in the study, with 30 patients in both groups eligible for the study. The patients were randomly divided into 2 groups. The randomisation in study was performed by using the closed envelope method. The TAP block was applied to Group I(Group S). The Group II(Group C) was patients who are not performed a block, and was taken as the control group. After all patients were taken to the operating table, ECG, non-invazive blood pressure, pulse oximetry and saturation monitoring were performed as the standard of ASA. During induction, 3mg/kg propofol, 1mg/kg fentanyl and 0.8 mg/ kg rocuronium were administered to all patients, then they were ventilated with 100% oxygen for 5 minutes and intubated with an appropriate intubation tube. After intubation in Grup S applied TAP block, the patients were covered with a sterile cleaned area, the transversus abdominis plane is visualized by placing the linear probe between the costal edge and the iliac wing, on the outer part of the abdominal wall, with a portable ultrasound device on the abdominal wall of the patients on the side to be repaired, and the external oblique muscle with the help of a 50 mm block needle. 0.25 % bupivacaine 0.5 ml/ kg maximum 20 ml was injected between the internal oblique and transverse muscles with in-plane tecnique. On the other hand, no blocks were applied to The Group C , and was taken as the control group. Anesthesia was maintained with 2% sevoflurane and 50% oxygen in air. Intravenous fluid maintenance was provied with isotonic-balanced electrolyte solution at 10 ml/kg/hour in both group. A maximum of 3 mg of morphine 50mcg/kg intravenously was given to all patients intraoperatively for analgesic purposes. At the end of the surgery, the patients were extubated under appropriate conditions.

Evaluation of postoperative pain; It was planned to be performed by a physician or a pain staff who did not perform the block, first in the postoperative recovery room and then in the ward, using The Wong-Baker Faces Pain Rating Scale (FACES Scale). The primary outcome of the study is The Wong-Baker Faces Pain Rating Scale (FACES Scale) scores of the patients, and the secondary outcomes are; time and amount of first additional rescue analgesic requirement, systolic-diastolic-mean arterial pressures, heart rate peaks and parental satisfaction scores. With predetermined time points; Postoperative baseline 0, 1st, 3rd, 6th, 12th and 24th hours of the patients' is The Wong-Baker FACE Scale scores, rescue analgesic totally amount, systolic-diastolic-mean arterial pressures, peak heart rates, and possible complications such as nausea and vomiting were recorded in both groups. Parental satisfaction levels were recorded on a numerical scale from 1 to 10 (1: lowest satisfaction, 10: highest satisfaction). If The Wong-Baker FACE Scale scores > 4, acetaminophen 10 mg/kg IV was planned to be administered as an additional rescue analgesic in the ward. In this study, power analysis was performed after the analysis results. Sample size was calculated by power analysis based on data from a previous study (12). In this study, researchers; They compared the analgesic effectiveness of the patients who applied TAP block and the placebo-control group in the first 48 hours postoperatively in a total of 60 patients who underwent pediatric appendectomy, and revealed that Tap block provided superior analgesia compared to the placebo group. Power estimation analysis suggested that add 30 individuals to each group and the power of the test was found to be p= 0.9035. The error level was taken as 0.05. In this study, when α= 0.05 β= 0.10 1-β = 0.90.

ELIGIBILITY:
Inclusion Criteria:

Those who have had surgery for acute appendicitis ASA status I-II

Exclusion Criteria:

ASA III-IV Perforated appendectomies Laparoscopic cases Patients allergic to local anesthetic drugs. Bleeding diathesis Skin infection at the needle entry site Those who refused to participate in the study.

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Patients aged between 5 and 16 years who were scheduled for elective open appendectomy surgery under general anesthesia were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2022-10-15 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Effect on pain score | At 0, 1, 3, 6, 12 and 24 hours after surgery
  Wong-Baker FACE Scale scores of patients were measured at 0, 1, 3, 6, 12 and 24 hours after surgery. Wong Baker FACE scale score will be scored as 10 at the highest and 1 at the lowest. The Turkish version has been adjusted for pediatric patients.

SECONDARY OUTCOMES:
Rescue analgesic consumption | At 0, 1, 3, 6, 12 and 24 hours after surgery
  If the Wong-Baker FACE Scale score was > 4, 10 mg/kg IV paracetamol was planned to be administered as additional rescue analgesia in the ward.

OTHER OUTCOMES:
Parental satisfaction levels | At 0, 1, 3, 6, 12 and 24 hours after surgery
  Parental satisfaction levels were recorded on a numerical scale from 1 to 10 (1: lowest satisfaction, 10: highest satisfaction).

CONTACTS AND LOCATIONS:
Locations (1):
- Arnavutkoy State Hospital, Istanbul, Arnavutkoy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mai CL, Young MJ, Quraishi SA. Clinical implications of the transversus abdominis plane block in pediatric anesthesia. Paediatr Anaesth. 2012 Sep;22(9):831-40. doi: 10.1111/j.1460-9592.2012.03916.x. PMID 22834467
- [Background] Seyedhejazi M, Motarabbesoun S, Eslampoor Y, Taghizadieh N, Hazhir N. Appendectomy Pain Control by Transversus Abdominis Plane (TAP) Block in Children. Anesth Pain Med. 2019 Feb 20;9(1):e83975. doi: 10.5812/aapm.83975. eCollection 2019 Feb. PMID 30881907
- [Background] Carney J, Finnerty O, Rauf J, Curley G, McDonnell JG, Laffey JG. Ipsilateral transversus abdominis plane block provides effective analgesia after appendectomy in children: a randomized controlled trial. Anesth Analg. 2010 Oct;111(4):998-1003. doi: 10.1213/ANE.0b013e3181ee7bba. Epub 2010 Aug 27. PMID 20802056
- [Background] Niraj G, Searle A, Mathews M, Misra V, Baban M, Kiani S, Wong M. Analgesic efficacy of ultrasound-guided transversus abdominis plane block in patients undergoing open appendicectomy. Br J Anaesth. 2009 Oct;103(4):601-5. doi: 10.1093/bja/aep175. Epub 2009 Jun 26. PMID 19561014